CLINICAL TRIAL: NCT06206161
Title: Testing Scalable, Broad-Reach School-Based Brief Interventions for Alcohol Use
Brief Title: Optimizing and Advancing SBIRT in Schools
Acronym: OASIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: C4 Innovations, LLC (Unknown); Harvard University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023P000998; AU-2022C1-26355 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Drinking; Adolescent Substance Use; Risk Behavior, Health
Keywords: Alcohol Use; Screening, Brief Intervention, Referral to Treatment (SBIRT); Prevention; Expanded Workforce
MeSH Terms: conditions — Underage Drinking; Health Risk Behaviors; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IPO, CLIN (Active Comparator): Standard brief intervention eligibility criteria involving indicated prevention (i.e., brief interventions delivered to high-risk drinkers only). BIs delivered by standard SBIRT workforce involving school nursing or clinical staff.
  Interventions: Behavioral: Indicated Prevention, Clinical Staff
- IPO, CLIN+PARA (Experimental): Standard brief intervention eligibility criteria involving indicated prevention (i.e., brief interventions delivered to high-risk drinkers only). BIs delivered by expanded SBIRT workforce involving school nursing or clinical staff and trained paraprofessionals.
  Interventions: Behavioral: Indicated Prevention, Clinical Staff; Behavioral: Expanded Paraprofessional Workforce
- SIP, CLIN (Experimental): Expanded brief intervention eligibility criteria involving selective prevention in addition to indicated prevention (i.e., brief interventions delivered to current drinkers with and without risky alcohol use). BIs delivered by standard SBIRT workforce involving school nursing or clinical staff.
  Interventions: Behavioral: Indicated Prevention, Clinical Staff; Behavioral: Selective Prevention
- SIP, CLIN+PARA (Experimental): Expanded brief intervention eligibility criteria involving selective prevention in addition to indicated prevention (i.e., brief interventions delivered to current drinkers with and without risky alcohol use). BIs delivered by expanded SBIRT workforce involving school nursing or clinical staff and trained paraprofessionals.
  Interventions: Behavioral: Indicated Prevention, Clinical Staff; Behavioral: Selective Prevention; Behavioral: Expanded Paraprofessional Workforce

INTERVENTIONS:
Behavioral: Indicated Prevention, Clinical Staff — Standard brief intervention eligibility criteria involving indicated prevention (i.e., brief interventions delivered to high-risk drinkers only). BIs delivered by standard SBIRT workforce involving school nursing or clinical staff.
Behavioral: Selective Prevention — Expanded brief intervention eligibility criteria involving selective prevention in addition to indicated prevention (i.e., brief interventions delivered to current drinkers with and without risky alcohol use).
  Arms: SIP, CLIN; SIP, CLIN+PARA
Behavioral: Expanded Paraprofessional Workforce — Brief interventions delivered by expanded SBIRT workforce involving school nursing or clinical staff and trained paraprofessionals.
  Arms: IPO, CLIN+PARA; SIP, CLIN+PARA

SUMMARY:
The goal of this clinical trial is to establish whether brief interventions for alcohol use can be delivered in schools for both indicated prevention and selected prevention, determine if an expanded workforce is an effective model for screening, brief intervention, and referral to treatment (SBIRT) delivery in schools, and explore whether brief intervention effectiveness is comparable in minoritized versus non-minoritized adolescents.

Participants will be students at high schools across Massachusetts. High schools will be randomized to one of four intervention groups. Participants will complete a baseline survey prior to their school-wide screening for SBIRT, and then will complete four follow-up surveys over two years.

DETAILED DESCRIPTION:
Massachusetts is the only state in the United States that mandates annual Screening, Brief Intervention and Referral to Treatment (SBIRT) assessments in public middle and high schools. SBIRT includes administering a validated screening instrument (CRAFFT + N) to all students in a single grade and then, based on responses on the screen, delivering a brief intervention (BI) to increase motivation to reduce substance use. While SBIRT represents a positive step in utilizing schools to enhance youth health, current BI implementation has limitations. Firstly, robust BIs primarily target youth already engaged in risky drinking, potentially neglecting those in need of early intervention. Secondly, relying on nursing and clinical staff for BI delivery strains an already burdened workforce. Exploring the inclusion of paraprofessionals, such as peers and mentors, can alleviate this burden and expand outreach. Lastly, there's a gap in ensuring the effectiveness of BIs for minoritized youth who face greater risks of alcohol-related issues.

The purpose of this study is to: 1) Establish whether BIs can be delivered in schools for both indicated prevention - i.e., for high-risk adolescents who already have signs of alcohol problems-and selective prevention - i.e., for moderate-risk adolescents prior to the emergence of problems from use. Public health recommendations for substance use prevention unequivocally advocate for the delivery of interventions as early in the use trajectory as possible. The entire foundation of SBIRT is predicated on this notion. However, BIs have largely been tested only in risky drinkers. (2) Determining if an expanded workforce is an effective model for SBIRT delivery in schools. While SBIRT has historically relied on nurse and clinician facilitation, there is a significant behavioral health workforce shortage that may hamper long-term sustainability, result in incomplete access for low-to-moderate-risk students, and magnify inequities in under-resourced schools. Other behavioral health disciplines have found great promise in embedding trained paraprofessionals into clinical workflow, but this has not been examined for school-based SBIRT. (3) Exploring whether BI effectiveness is comparable in minoritized vs non-minoritized adolescents. While preliminary studies have shown SBIRT to improve system equity and efficiency, this does not always translate to consistent screening and culturally responsive care. This study will explicitly seek to explore heterogeneity in BI effectiveness and use this to inform the development of more equitable, culturally responsive interventions to reduce disparities and increase access.

To address these scientific gaps, the research team aims to test the effects of (1) standard vs expanded criteria for BI eligibility (IPO [TAU] vs. SIP) and (2) standard vs expanded SBIRT workforce (CLIN [TAU] vs. CLIN+PARA) on alcohol, other substance use, and mental health outcomes over 24 months. Investigators will conduct 2x2 analyses of these effects in a cluster randomized trial of 40 high schools in Massachusetts, in which the investigators will survey ~21,000 10th-grade adolescent students over two years and analyze data from a conservative estimate of ~1,900 with past-year alcohol use. The investigators will also enroll an estimated 19,100 students with never or less than past year alcohol use to explore the impact of the target BI intervention strategies (BI eligibility criteria and SBIRT workforce) on initiation of alcohol use and progression among those with low-risk (i.e., never or less than past-year) alcohol use. Participants will be assessed prior to SBIRT screening and then approximately every six months over a 24-month follow-up period. The length of this follow-up period will allow assessment of alcohol use across critical developmental windows during which progression is most common (i.e., 10th through 12th grade, inclusive of two summer vacations). Investigators hypothesize that BIs delivered with expanded eligibility criteria and an expanded workforce, i.e., SIP and CLIN+PARA, will be associated with better substance use and mental health outcomes across the four post-baseline sessions because more proactive prevention will provide skills to more students to buffer against the risk of progression earlier in the substance use trajectory. An expanded workforce will have more time to deliver BIs, follow-up, and referrals, resulting in greater capacity for higher doses of BIs in schools. The investigators suggest that expanded eligibility and an expanded workforce are best deployed in tandem because more inclusive prevention targets (i.e., via SIP) will inevitably result in larger caseloads, and paraprofessionals with dedicated time can help mitigate this burden.

The qualitative aims for this study will be to explore barriers to implementing the studied BI approaches and heterogeneity in BI effects in REM, LBGTQ+, and ELL participants. To accomplish the first part of this aim, investigators will conduct individual semi-structured interviews with school staff and paraprofessionals to assess beliefs around school-based substance use prevention as well as structural factors that may impact access to supports, effectiveness, and sustainability. The study team will also conduct 80 individual interviews with students enrolled in the longitudinal study. Interview participants will be samples by treatment arm (CLIN+PARA versus CLIN; IPO versus SIP), substance use status (low/moderate versus high), and minority status (REM, LGBTQIA+, ELL).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a participating high school and in the grade scheduled to receive SBIRT

Exclusion Criteria:

* Passive consent declined by parent/guardian through the opt-out model

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21000 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Past 30-day alcohol use frequency | 6, 12, 18, and 24 months
  Past 30-day alcohol use frequency (number of days) will be assessed via self-report questions from the Monitoring the Future (MTF) survey.
Past 30-day cannabis use frequency | 6, 12, 18, and 24 months
  Past 30-day cannabis use frequency (number of days) will be assessed via self-report questions from the Monitoring the Future (MTF) survey.
Past 30-day nicotine use frequency | 6, 12, 18, and 24 months
  Past 30-day nicotine use frequency (number of days) will be assessed via self-report questions from the Monitoring the Future (MTF) survey.

SECONDARY OUTCOMES:
Number of Alcohol Problems | 6, 12, 18, and 24 months
  Number of alcohol-related problems will be assessed using the Alcohol Use Disorders Identification Test (AUDIT). The AUDIT has a range from 0 to 40, with higher scores indicating more alcohol-related problems. Scores of 5 or greater indicate hazardous drinking in adolescents.
Binge Drinking Episode Frequency | 6, 12, 18, and 24 months
  Binge drinking episode frequency will be assessed via self-report questions from the Monitoring the Future (MTF) survey. Assessments will use a developmentally-scaled definition of binge drinking defined as ≥4 drinks and ≥3 drinks in two hours for 14-15 year old males and females, respectively, and ≥5 drinks and ≥3 drinks in two hours for 16-17 year old males and females, respectively.
Past 2-week depression symptoms | 6, 12, 18, and 24 months
  Depression symptoms will be assessed using the Depression subscale of the Patient Health Questionnaire-4 (PHQ-4). This subscale ranges from 0-6, with higher scores indicating greater symptoms burden. Scores of 3 or greater on the depression subscale of the PHQ-4 are suggestive of potential cases of major depression or other depressive disorders.
Past-year thoughts of suicide | 12 and 24 months
  Past-year thoughts of suicide will be assessed using a self-report measure. The measure will query about past-year passive suicidal ideation, active suicidal ideation, suicidal preparatory acts and behavior, and non-suicidal self-injury. Binary (yes/no) response options will be provided.
Past 2-week anxiety symptoms | 6, 12, 18, and 24 months
  Anxiety symptoms will be assessed using the Depression subscale of the Patient Health Questionnaire-4 (PHQ-4). This subscale ranges from 0-6, with higher scores indicating greater symptoms burden. Scores of 3 or greater on the Anxiety subscale of the PHQ-4 are suggestive of potential cases of generalized anxiety, panic, social anxiety, and posttraumatic stress disorders.
Number of Referrals | 6, 12, 18, and 24 months
  The number of referrals to follow-up support services will be assessed via self-report questionnaire. Subjects will be asked whether they have met with someone at school (not including a friend or another student) since their last assessment about mental health and substance use (yes/no). If yes, they will receive additional questions to understand the role of the person/people they met with, topics addressed, duration and intensity of the encounter(s), and perceived helpfulness of the support received.

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The full data package, which includes the de-identified analyzable data set, full protocol, metadata, data dictionary, full statistical analysis plan (including all amendments and all documentation for additional work processes), and analytic code, will be shared with a controlled-access, PCORI-designated repository as outlined in the PCORI Policy for Data Management and Data Sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 90 days of submission of the draft final research report and will be maintained in the repository for at least 7 years.
Access Criteria: Investigators seeking access to the data from this PCORI-funded trial will need to complete and submit a data access request to the PCORI-designated repository. The repository will review requests based on the qualifications of the investigators and scientific merit. If the request is approved, the requestor's institution will need to enter into a data use agreement with the PCORI-designated repository with will specify terms and conditions for data use.